CLINICAL TRIAL: NCT06412159
Title: Intra-oral Digital Evaluation of Fit Accuracy for Removable Partial Denture Frameworks Fabricated by Selective Laser Melting Using 2 Different Impression Techniques. Within Subjected Study
Brief Title: Digital Evaluation of Accuracy for Removable Partial Denture Frameworks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Ragheb, associate professor, Kafrelsheikh University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-130
Record Dates: First submitted 2024-05-03; First posted 2024-05-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Denture; Partial
Keywords: partial denture; intra oral; digital evaluation; accuracy; selective laser melting

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selective laser melting removable partial denture frameworks fabricated by conventional technique (Other): selective laser melting removable partial denture frameworks fabricated by conventional technique
  Interventions: Other: Selective laser melting framework was fabricated using completely digital workflow
- selective laser melting framework was fabricated using completely digital workflow (Other): selective laser melting framework was fabricated using completely digital workflow
  Interventions: Other: Selective laser melting framework was fabricated using completely digital workflow

INTERVENTIONS:
Other: Selective laser melting framework was fabricated using completely digital workflow — completely digital work flow Conventional technique versus complete digital technique

SUMMARY:
Purpose:Within subject study aim to compare the overall accuracy and fit of different components for mandibular metallic removable partial denture (RPD) frameworks fabricated by selective laser melting using combined analog-digital, and fully digital impression techniques.

Material and methods. Two RPD frameworks were fabricated for each of the 24 participants using each of the 2 techniques of the 24 participants enrolled, were of mandibular Kennedy class I, the first technique was the combined analog-digital workflow had the analog steps include: a physical impression was made using polyvinyl siloxane, stone casts were made, then the stone cast was scanned with a laboratory scanner to generate a digital cast. The 3Shape CAD software was then used to design a digital RPD, which was fabricated from a cobalt-chroumum alloy by selective laser melting. The second technique was fully digital where an intraoral digital scanner was used to make a definitive scan, which was sent to the 3Shape software for digitally designing the RPD framework and subsequent selective laser melting for fabrication. For both frameworks in the same participant, the same design was used for consistency. To assess the accuracy of fit, based on STL data analysis (intra-oral digital superimposition evaluation), a color map was constructed using non metrology software, and overall fit accuracy and the misfit (distance between each framework component and the reference intra-oral scan) were measured at rest, guiding plane and lingual plate areas.

DETAILED DESCRIPTION:
Twenty four mandibular bilateral partially edentulous participants aged from 50 to 65 years having mandibular Class I Kennedy classification were selected randomly from the outpatient clinic of the prosthodontic department. The clinical study was explained to the patients and they accept it and an informed consent were signed by all them

For each patient, two different cobalt chromium removable partial denture frameworks were constructed; the first one was fabricated using combined analog-digital workflow (group 1) and the other framework was fabricated using completely digital workflow (group 2) and comparing them through evaluation of:

1. Over all accuracy
2. Accuracy of fit of occlusal rests, major connector, Guiding plane/plate relation and retentive terminal of I bar clasp.

Two techniques were used to fabricate 48 RPD frameworks in total. Fabrication of cobalt chromium removable partial denture framework using combined analog-digital workflow (group 1)

The Removable partial denture frameworks for group 1 were fabricated as follow:

The first technique was a combined analog-digital technique, in which a physical definitive impression was made and a stone cast was fabricated. a physical impression was made using polyvinyl siloxane impression material. , and a stone cast was poured using Type IV stone . In an edentulous area, border molding was first accomplished using a green modeling plastic impression compound . The impression and stone cast were evaluated critically to ensure quality. The stone cast was then scanned using a laboratory scanner to produce a virtual 3D master model. The 3Shape CAD software was used to design a digital RPD . The RPD framework was designed with an lingual plate mandibular major connector, I bar retentive clasps on the first premolars.

The definitive STL design file was then sent to the Dental Laboratory, to be selective laser melted in Co-Cr alloy.

The Overall fit accuracy and the misfit at some areas where the accuracy measurement was performed, included: The rest/rest seat areas of right and left premolars , the right and left guide plane/plate area , the mandibular major connector area including the superior border of lingual plate area and retentive terminal of I bar clasp.

All measurements were made by a single investigator and were repeated five times. The average error of measurement was approximately 0.002 mm. As a basis for our evaluation of misfit, a distance of 0 to 0.05 mm was considered close contact (no gap), and a distance of 0.05 to 0.31 mm was defined as clinically acceptable fit.

ELIGIBILITY:
Inclusion Criteria:

* mandibular Class I Kennedy classification were selected randomly from the outpatient clinic of the prosthodontic department

Exclusion Criteria:

* other classes of removable partial denture maxillary partially edentulous patients

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Intra-oral digital Evaluation of fit accuracy for removable partial denture frameworks | immediately after insertion of removable partial denture frame work
  Intra-oral digital Accuracy of fit evaluation between frame works by using medit compare software to exclude the value of point difference in different area at occlusal rest major connector

CONTACTS AND LOCATIONS:
Locations (1):
- Nourhan Ragheb, Kafr Elsheikh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elgamal M, Ibrahim AM, Fadl BT, Ragheb NA. Accuracy assessment of removable partial denture frameworks fabricated by selective laser melting using two different workflows: A cross-over clinical study. BMC Oral Health. 2025 May 28;25(1):824. doi: 10.1186/s12903-025-06214-9. PMID 40437453